CLINICAL TRIAL: NCT00283621
Title: A Pilot Study of Aranesp (Darbepoetin Alfa) and Pegfilgrastim (Neulasta) in Patients With Sarcoma Receiving Adriamycin and Ifosfamide
Brief Title: Aranesp and Neulasta in Patients With Sarcoma Receiving Adriamycin and Ifosfamide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ID02-326
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Sarcoma
Keywords: Aranesp; Darbepoetin Alfa; Pegfilgrastim; Neulasta; Sarcoma; Adriamycin; Doxorubicin Hydrocholoride; Adriamycin PFS; Adriamycin RDF; Ifosfamide
MeSH Terms: conditions — Sarcoma | interventions — Darbepoetin alfa; pegfilgrastim; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Growth Factors + Adriamycin/Ifosfamide (Experimental): Growth Factors = Aranesp (Darbepoetin Alfa) and Pegfilgrastim (Neulasta)
  Interventions: Drug: Aranesp (darbepoetin alfa); Drug: Neulasta (pegfilgrastim); Drug: Adriamycin; Drug: Ifosfamide

INTERVENTIONS:
Drug: Aranesp (darbepoetin alfa)
Drug: Neulasta (pegfilgrastim)
Drug: Adriamycin
  Other Names: Doxorubicin Hydrocholoride; Adriamycin PFS; Adriamycin RDF
Drug: Ifosfamide
  Other Names: Ifex

SUMMARY:
To determine the percentage of patients and number of cycles in which a packed red blood cell transfusion was administered due to anemia and in which antibiotics were administered due to neutropenic fever.

DETAILED DESCRIPTION:
The use of hematopoietic growth factors have been shown to reduce neutropenic complications and red cell transfusion requirements associated with chemotherapy. This trial will study the combination of pegfilgrastim and darbepoetin alfa administered once per cycle of chemotherapy. Prior experience with growth factors in this setting provides historical data for comparison of safety and activity of these newer longer acting growth factors in reducing the incidence of febrile neutropenia requiring antibiotics and anemia requiring transfusions. The once dosing per cycle would simplify the patient management and would improve patient convenience and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sarcoma which is locally advanced, at high risk for relapsed or metastatic for whom treatment with AI is indicated
* Must be between 18-65 years of age
* Women of childbearing potential should use effective contraceptive measures
* Adequate hematologic, renal, and hepatic functions
* Karnofsky performance status above or equal to 80

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with comorbid condition which renders patients at high risk of treatment complication
* Patients with metastatic disease to CNS
* Patients with significant cardiac abnormalities
* History of seizure disorder in the past 5 years
* Patient has received any packed red blood cell transfusion within 2 weeks before study entry
* Prior surgery or radiation therapy within 2 weeks of study entry
* History of prior chemotherapy for sarcomas
* Iron deficiency
* Hypersensitivity to E.coli derived products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-06-02 (Actual); Primary Completion 2006-04-12 (Actual); Study Completion 2006-04-12 (Actual)

PRIMARY OUTCOMES:
CBC diff/platelet counts | Monitored at least twice a week and daily during severe myelosuppression.
Iron Stores | Blood drawn at baseline during cycle 3 and at the end of study.
Peripheral blood and bone marrows | Performed at baseline and post treatment.

SECONDARY OUTCOMES:
Neurocognitive functions and Symptom burden assessment | Assessed at baseline, after 3 cycles of treatment and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, M.D., Principal Investigator — UT MDAnderson Cancer Center
Locations (1):
- UT MDAnderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org